CLINICAL TRIAL: NCT03078998
Title: The Investigation of Effectiveness of Leap Motion Based Exercises in Upper Extremity Rehabilitation of The Children
Brief Title: Leap Motion Based Exercises in Upper Extremity Rehabilitation of The Children
Acronym: LMBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ela Tarakci, Assoc.Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 108400987275
Record Dates: First submitted 2017-03-02; First posted 2017-03-14 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Rehabilitation; Physical Therapy
Keywords: Juvenile Idiopathic Arthritis; Cerebral Palsy; Obstetric Brachial Plexus Palsy; Human Computer Interaction; Leap Motion; Video Game Based Rehabilitation
MeSH Terms: conditions — Arthritis, Juvenile; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Juvenile idiopathic Arthritis (Experimental)
  Interventions: Device: Leap Motion Based Exercises
- Obstetric Brachial Plexus Palsy (Experimental)
  Interventions: Device: Leap Motion Based Exercises
- Cerebral Palsy (Experimental)
  Interventions: Device: Leap Motion Based Exercises

INTERVENTIONS:
Device: Leap Motion Based Exercises — Game based exercise

SUMMARY:
Juvenile Idiopathic Arthritis (JIA), Cerebral Palsy (CP), and Obstetric Brachial Plexus Injury (OBPI) are the most common disorders that cause upper extremity impairments in children. Depending on the underlying pathologies, the common symptoms of these disorders are the limitations of the upper extremity joint movement angles, muscle imbalance and the functional limitations caused by the contracture due to these problems. Daily life activities such as feeding, personal care, and self mobility activities that use upper extremity are commonly limited with these children. Physical rehabilitation is mostly used to address these problems. However, the process of rehabilitation is difficult and lengthy. In addition, most of the time, classical rehabilitation is discouraging for many young patients. Employment of digital technology has been gaining momentum in addressing the above rehabilitation problems among the medical professionals.

By utilizing exciting new sensor technologies, such as Microsoft Kinect, Nintendo Wii and Leap Motion, practical game based rehabilitation applications have been becoming popular. Video Based Games (VBG) that adopt the these technologies as Human Computer Interaction (HCI) interfaces are recently used successfully for the task of rehabilitation. The Leap Motion device, one of the new examples of these technologies, has a very small form factor. It includes two near infrared stereoscopic cameras to capture hand images of patients to produce 3 Dimensional (3D) positions of hand joints at a very fast rate with a sufficient positional precision.

There have been examples that use motion sensor based VBG's for the rehabilitation of different types of patient groups. Compared to classical rehabilitation practices, these applications provide many advantages such as ease of use, repeatableness, and instantaneous measurable feedback. In addition, the young patients involved in these applications demonstrated willingness to participate in these activities and they showed considerable progress in upper extremity rehabilitation. However, these VBG's were mostly developed for general public and it was often suggested to develop VBG's for the specific task of upper extremity rehabilitation of children. It is known that upper extremity specific VBG's and their applications are very limited both at the global and domestic levels.

With this project, we plan to design and develop specialized Leap Motion based VBG's for the children diagnosed with JIA, CP, and OBPI. These VBG's will be designed to be easy to use and motivating for the children. They will automatically lead the patients to correct hand exercises and they will provide mechanisms for online performance measurements of the patients. The performance results from the patients will be compared with the results from the classical rehabilitation applications by the standards of The International Classification of Functioning (ICF). These games will provide complete Turkish language support for the extended national dissemination of the project outputs.

The proposed project is inherently a multi disciplinary work that requires very close interaction of phisiotherapists, software experts, and HCI specialists and efficient application of the these games for the patients. There will be specialized games for each disorder. These games will utilize the outputs from the Leap Motion device that will produce 3D hand joint positions and joint angles. Realistic animations of hand and virtual environments will provide a motivating exercise game platform for the patients.The performance measurements of the patients will be repeated for each game session. There will be game parameters for the game duration, difficulty level, and hand joints in focus. The game hand movements will reflect daily life activities for the rehabilitation purposes which would make our games different from the general public games. The project findings at end of the project on best game usage frequency and durations, the effectiveness of the designed VBG's and other results will be shared with the scientific community through publications and seminars.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile idiopathic Arthritis, Cerebral Palsy, Obstetric Brachial Plexus Palsy have been diagnosed,
* 5-17 years of age,
* In the last 6 months, no other treatment, such as Botarinium Toxin (BOTOX) injection, intraarticular injection, surgery, which can affect extremity rehabilitation,
* Upper extremity Modified Ashworth Scale (0), (1), (1+) for children wtih Cerebral palsy
* Having the ability to adapt to exercises

Exclusion Criteria:

* Diagnosed cardiac or orthopedic disorders that may interfere with the application of evaluation methods,
* Having a mental problem

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Jebsen Taylor Hand Function Test | 8 weeks

SECONDARY OUTCOMES:
Nine Hole Peg Test | 8 weeks
Childhood Health Assessment Questionnaire | 8 weeks
Duruoz Hand Index | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ela Tarakci, Principal Investigator — Istanbul University; Nilay Arman, Study Director — Istanbul University; Devrim Tarakci, Study Director — Medipol University; Yusuf Sinan Akgul, Study Chair — Gebze Institute of High Technology

IPD SHARING:
Plan to Share IPD: No